CLINICAL TRIAL: NCT06689111
Title: Investigation of Whether the Presence of the Typical LBBB- Mechanical Stimulation Pattern - Documented Through 2DSE (Two-dimensional Strain Echocardiography) - is Associated With Increased Rates of Acute Improvement in Global Myocardial Work Efficiency (GWE) Compared to the Absence of This Activation Pattern, in Patients in Need of Device Implantation for Cardiac Resynchronization Therapy in Whom LBBp is Chosen Compared to the Classic Biventricular Pacing Method
Brief Title: Correlation of Typical LBBB Mechanical Activation Pattern by 2D Strain Echocardiography With Acute GWE Improvement in Patients Receiving LBBp or Conventional BiVp for Cardiac Resynchronization Therapy (Echo LBBp)
Acronym: ECHO-LBBp
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Patras (Other)
Collaborators: University General Hospital of Heraklion (Other); Ippokrateio General Hospital of Thessaloniki (Other); Onassis Cardiac Surgery Centre (Other); Alexandra Hospital, Athens, Greece (Other); Korgialenio-Benakio Red Cross Hospital (Other); Ippokration General Hospital (Other)
Responsible Party: Principal Investigator, Georgios Leventopoulos, Principal Investigator, University Hospital of Patras
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 337/23.05.2024
Record Dates: First submitted 2024-10-31; First posted 2024-11-14 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure With Reduced Ejection Fraction (HFrEF)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Left Bundle branch Pacing (Experimental): Implantation of a left bundle branch lead via sheath, to perform left bundle branch pacing
  Interventions: Device: Left bundle branch pacing lead
- Conventional Bi- Ventricular pacing (Active Comparator): Conventional resynchronization therapy using a vein through coronary sinus
  Interventions: Device: CRT with the standard method through cs

INTERVENTIONS:
Device: Left bundle branch pacing lead — Use of LBBp Vs the standard method of BiVp in resynchronization therapy
  Arms: Left Bundle branch Pacing
Device: CRT with the standard method through cs — standard CRT procedure
  Arms: Conventional Bi- Ventricular pacing

SUMMARY:
The present study is a multicenter interventional non randomised study in patients requiring an implantable device for cardiac resynchronization therapy. Its primary objective is to investigate whether the presence of a specific echocardiographic contraction pattern before implantation is associated with increased rates of acute improvement in myocardial function (as measured by an ultrasound) and to compare the improvement in two groups of patients based on the type of pacing (biventricular or left-sided pacing)

DETAILED DESCRIPTION:
There is now sufficient evidence that the presence of typical LBBB mechanical stimulation on 2D Strain Echocardiography - and not simply the presence of electrocardiographic criteria - is associated with increased rates of adequate response to resynchronization therapy with implantable CRT relative to patients who met electrocardiographic criteria for LBBB without however, the typical stimulation pattern documented echocardiographically.

Identification criteria of LBBB typical mechanical stimulation in 2DSE are :1) early shortening of at least 1 basal or mid-ventricular segment in the septal wall and early stretching in at least 1 basal or midventricular segment in the lateral wall, 2) early septal peak shortening (within the first 70% of the ejection phase), and 3) lateral wall peak shortening after aortic valve closure.

The absence of one of the three criteria categorizes the patient in the group of atypical LBBB stimulation pattern.

Along with the development of the newest non-invasive imaging methods using ultrasound, the calculation of myocardial work (Myocardial Work) as well as the calculation of GWW (Global Wasted Work), GCW (Global Constructive Work) and GWE (Global Work Efficiency) is possible and can be used as a way of assessing myocardial function, the response to administered treatment (e.g. resynchronization therapy) as well as in the search for patients with the most likely response to a possible treatment.

The purpose of the study is to investigate which patients are most likely to benefit from LBBP pacing. Classic biventricular pacing will be compared with LBB pacing in patients requiring resynchronization with LVEF < 35%. At the same time, the presence or not of a typical LBBB- pattern of mechanical stimulation will be evaluated - documented through 2DSE (Two-dimensional strain echocardiography). - The immediate improvement of GWE in patients with succeeded LBB pacing - as documented by measurements in the electrophysiological laboratory- will be compared to the group of patients with the classical method of biventricular pacing (BiVp) as well as the correlation of the presence of the sonographic pattern of LBBB stimulation compared to the group of patients who do not present this mechanical activation pattern in ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* >18 years < 90 years
* Patients with a documented indication for resynchronization therapy [symptomatic patients despite optimal medication, HFrEF (EF<35%), LBBB QRS morphology]
* COMPLETE LBBB (LBBB defined as QRS>130msec, wide "notched or slurred" R wave in leads I, aVL, V5, V6 and occasional RS pattern in V5, V6, absence of Q waves in leads I, V5 and V6 but in lead aVL narrow Q wave may be present in the absence of myocardial pathology, R peak time >60ms in leads V5 and V6 but normal in leads V1, V2, V3 when small R's are discernible in precardial leads, ST and T usually opposite to QRS direction)
* Patients with ntraventricular septum diameter >8 mm
* Written informed consent

Exclusion Criteria:

* Patients with RBBB or atypical LBBB QRS morphology
* Patients eligible for an upgrade procedure (already carring a PM or ICD)
* Patients with hypertrophic cardiomyopathy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
GWE IMPROVEMENT | Comparison in the acute phase after implantation (first to second day after the implantation))
  Echocardiographic dyssynchrony index change, as expressed with Global Left Ventricular Myocardial Work Efficiency (GWE) (%) Change of myocardial work after LBBP/CRT implantation (correlation before and after)* and comparison in four groups based on the method of resynchronization (LBBp and BiVP) and ultrasound findings: a) Echo pattern typical LBBB b) Echo pattern atypical LBBB

SECONDARY OUTCOMES:
Successful LBB pacing | first day after the procedure
  These include the presentation of R' in V1 and at least on of the following:
  1. Threshold test: the transition from nonselective LBBP (NS-LBBP) to S-LBBP
  2. V6RWPT< 80ms
  3. V6-V1 inter-peak interval >44ms
  4. Potential- V6RWPT =stim-V6RWPT (+/-10ms)
  5. QRS transition ns - LBBB to s-LBBB by programmed stimulation S1S2
Complications associated with pacemaker implantation | first day after the procedure
  General device related complications: pneumothorax, hemothorax, infection, tamponade, hematoma, lead reoperation Specific complications associated with the left bundle branch pacing procedure: intraventricular septum rupture, septal perforator branch injury with subsequent myocardial infarction or lead displacement
Procedure and Fluroscopy time (min) | first day after the procedure
  Total procedure and fluroscopy time

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Patras, Pátrai, Greece, Greece